CLINICAL TRIAL: NCT00327249
Title: A Phase 1/2 Trial of Amplimexon® (Imexon, Inj.) for Patients With Previously Treated Multiple Myeloma
Brief Title: Safety and Efficacy Study of Imexon for Treatment of Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Evan Hersh, AmpliMed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP-007
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: imexon

SUMMARY:
AMP-007 is a Phase 1/2 study for the treatment of advanced, previously treated multiple myeloma. The first phase of the study is designed to determine a safe dose of imexon that can be given to patients with advanced, previously-treated multiple myeloma. The Phase 2 part of the study is designed to provide additional safety data and to gain an understanding of whether imexon can improve the outcome for patients with multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Advanced myeloma, with measurable disease as defined in the protocol.
* Prior treatment, at least 2 prior regimens are required. This may include prior treatment with investigational products.
* Able to perform the activities of daily living.
* Off prior therapy for at least 2-4 weeks depending on the drug.
* Blood counts and blood chemistries in or near normal range.
* If female, neither pregnant nor nursing.
* Willing to use contraceptives to prevent pregnancy.
* No other serious illnesses.
* No other active malignancy.
* No serious infections.
* No current other drug therapy for the myeloma except for steroid therapy under certain circumstances. Biphosphonate therapy is permitted.
* Prior radiation is permitted.

Exclusion Criteria:

* Use of corticosteroids for amyloid disorders, or high dose chronic steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximally tolerated dose of imexon in multiple myeloma patients
evaluate the toxicity of imexon
Preliminarily evaluate efficacy in terms of response and progression free survival.

SECONDARY OUTCOMES:
Evaluate biomarker responses.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigational Site 025, Little Rock, Arkansas
  - Investigational Site 008, Houston, Texas